CLINICAL TRIAL: NCT05216679
Title: Novel Stretching Device Versus Night Splints a Prospective, Randomized Study in the Effectiveness of Treating Plantar Fasciitis
Brief Title: Novel Stretching Device Versus Night Splints
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SAE Orthopedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tssfad1
Record Dates: First submitted 2022-01-03; First posted 2022-01-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-01

CONDITIONS: Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Main study (Experimental): This is the only arm of the study. It is a 6 week period where the participants will either be using night splints or the TESS device to treat their plantar fasciitis symptoms.
  Interventions: Device: Night splints; Device: Triceps Surae Stretching and Flexibility Assessment Device (TESS)

INTERVENTIONS:
Device: Night splints — A night splint is a brace the patient wears on their foot to keep it in a dorsiflexed position while they sleep. It is the first line treatment for plantar fasciitis.
Device: Triceps Surae Stretching and Flexibility Assessment Device (TESS) — The TESS device is a slant board with a bar added for balance that the participant will stand on in 5 minute intervals throughout the day to stretch their calves, and potentially treat their plantar fasciitis symptoms.

SUMMARY:
A set of 100 patients previously diagnosed with plantar fasciitis will be given initial questionnaires about their symptoms and randomly assigned either night splints or the novel calf stretching device. The participants will use each device for 6 weeks. At the end of those 6 weeks, they will return for a follow up questionnaire. The answers in the questionnaire will be analyzed to compare the effectiveness of night splints to calf stretching.

DETAILED DESCRIPTION:
The attached recruitment brochure will be distributed to physician's offices, and possibly placed as an ad in the newspaper. Potential participants will call the enclosed number and an appointment will be arranged to be evaluated at our research facility in Carterville, IL. During their initial evaluation which will take 30 minutes to 1 hour, each participant will complete medical history pertinent to plantar fasciitis and questionnaires regarding symptoms and physical activity. The research participants will then stand on the tssfad1 device for 5 to 10 minutes during which time their triceps surae flexibility will be assessed by measuring the distance from their heel to the platform at the 30-degree setting. Measurements for each foot will be taken with a distance sensor every 5 seconds for a 5 minute period.

The investigators will then use a random number generator program from www.random.org to generate a number between 1 and 100. Participants with an odd number will be assigned home use of standard night splints. Those with an even number will be provided with a TESS unit to be used at home a minimum of 5 minutes twice per day.

The participants will use their device for 6 weeks. They will receive a check in phone call at the 3 week mark of their participation.

Contact numbers will be given to each participant should they have any questions or concerns during the six-week interval. Each participant will be asked to maintain a daily log of their pain level on a visual analog scale and of their estimated time using each device.

Participant's random number will be used to link data in the study to the participant. The investigators will not be using patient identifiable information such as name, date of birth, medical record number, or other personal information for the record.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years and older
* diagnosis of plantar fasciitis
* ability to understand the purpose of the study
* ability to safely use the device they are assigned after education and return demonstration.

Exclusion Criteria:

* patients with ankle fusion or significant balance impairment which would prohibit safe use of the TESS device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-14 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who will attend follow up appointment and describe their symptoms and pain using a standard 0-10 pain chart. | 6 weeks
  The participant will return their device and fill out a questionnaire (the same as the original questionnaire from the first visit) that will ask them to describe their symptoms and pain levels using a standard 0-10 pain scale chart. The investigators will then use a Mixed ANCOVA statistical test to compare the effectiveness of the TESS device to night splints in symptom relief.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Davis', MD, Principal Investigator — SAE Orthopedics
Locations (1):
- SAE Orthopedics, Carterville, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
All data that underlie a publication will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available 6 months after study publication. Data will remain available indefinitely.
Access Criteria: Dr. Davis will review requests to access study data on a case by case basis. All deidentified data from this study has potential to be shared with other researchers. Requests can be made via email to james.m.davis1@siu.edu.